CLINICAL TRIAL: NCT06196697
Title: A Phase II, Single Arm, Single Center Study of Cadonilimab(AK104) in Combination With Ivonescimab(AK112) Plus Chemotherapy(SOX/XELOX) as First-line Treatment for Advanced Gastric (G) or Gastroesophageal Junction (GEJ) Cancer
Brief Title: AK104 in Combination With AK112 Plus Chemotherapy(SOX/XELOX) as First-line Treatment for Advanced G/GEJ Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yanqiao Zhang, professor, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-041
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: first-line treatment
MeSH Terms: interventions — XELOX; Oxaliplatin; Capecitabine; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104+AK112+SOX/XELOX (Experimental): Biological: Cadonilimab (AK104) 10mg/kg or 15mg/kg or 6mg/kg Q6W iv D8 (dose choosing depends on the outcome of the dose climb stage) Biological: Ivonescimab (AK112): 20mg/kg Q3W iv D1 Drug:SOX or XELOX SOX: Oxaliplatin (130 mg/m2 intravenous infusion for 2-6 hours on Day 1, Q3W,up to 6 cycles)+ Tegafur (40 mg/m2, p.o., Bid, Q3W, for day 1 to day 14 per cycle) XELOX: Oxaliplatin (130 mg/m2 intravenous infusion for 2-6 hours on Day 1, Q3W,up to 6 cycles)+Capecitabine(1000 mg/m2, p.o., Bid, Q3W, for day 1 to day 14 per cycle)
  Interventions: Biological: Cadonilimab; Biological: Ivonescimab; Drug: XELOX; Drug: SOX

INTERVENTIONS:
Biological: Cadonilimab — Subjects will receive AK104 by intravenous administration
  Other Names: AK104
Biological: Ivonescimab — Subjects will receive AK112 by intravenous administration
  Other Names: AK112
Drug: XELOX — Subjects will receive AK104 and AK112 in combination with XELOX(oxaliplatin and capecitabine)
  Other Names: oxaliplatin and capecitabine
Drug: SOX — Subjects will receive AK104 and AK112 in combination withSOX(oxaliplatin and Tegafur)
  Other Names: oxaliplatin and Tegafur

SUMMARY:
The goal of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, and anti-tumor activities of cadonilimab in combination with Ivonescimab plus chemotherapy as first-line therapy in adult subjects with HER2 negative、advanced or metastatic gastric (G) or gastroesophageal junction (GEJ) cancer.

DETAILED DESCRIPTION:
The study consists of a dose escalation and expansion phase to determine the recommended Phase 2 dose (RP2D) for AK104 in combination with AK112 and SOX/XELOX, and a dose confirmation phase which will further characterize the treatment of AK104 in combination at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent.
2. Imaging examination confirmed unresectable locally advanced or metastatic gastric cancer (GC) or gastroesophageal binding cancer (GEJC), and histopathologically confirmed adenocarcinoma, with at least one measurable tumor lesion (spiral CT or MR scan ≥10mm, gonorrhea The short diameter of sling is ≥15mm, which meets the RECIST 1.1 standard); the lesion that has received radiotherapy is not selected as the target lesion, unless the radiotherapy lesion is the only measurable lesion and is clearly advanced according to imaging judgment, it can be considered as the target lesion;
3. Subjects have not received prior systemic therapy for locally advanced or metastatic gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction. For subjects who have received prior neoadjuvant/adjuvant chemotherapy or chemoradiotherapy for curative intent, the time between disease progression and last treatment should be at least 6 months；
4. HER2 is negative. HER2 negative is defined as: IHC 0/1+, or IHC 2+ and FISH/ISH negative (HER2: CEP17 ratio <2). FISH can be replaced by locally available and accepted ISH methods (such as DISH);
5. The study allowed the inclusion of Subjects with gastric cancer with peritoneal metastasis (imaging results or ascites/abdominal lavage cytology test positive);
6. Expected survival period > 3 months;
7. ECOG score: 0-1;
8. All acute toxic reactions caused by previous anti-tumor treatment or surgery are relieved to level 0-1 (according to NCI CTCAE version 5.0) or to the level specified in the group/exclusion standard. Except for other toxicicies that researchers such as hair loss, fatigue and hearing damage believe do not pose a safety risk to the subjects;
9. Have good organ function (subsists are not allowed to receive blood transfusion or growth factor support treatment within 7 days before the first administration):

1) Absolute count of neutrophils ≥1.5×109/L; platelets ≥100×109/L; hemoglobulin ≥90g/L or 5.6mmol/L; 2) Total bilirubin ≤ 1.5 times the upper limit of normal value (ULN); ALT and AST ≤2.5×ULN, for liver metastasis subjects, ALT and AST ≤5×ULN; albumin ≥3.0g/dL (30g/L); 3) serum creatinine ≤1.5 ×ULN or calculated serum creatinine clearance ≥50mL/min (Cockcroft-Gault formula calculation).

4) Normal urine routine, or urine protein <2+; if urine protein ≥2+, the 24-hour urine protein quantity must be ≤1g; 5) Normal coagulation function, international standardization ratio (INR) ≤ 1.5×ULN, prothrombin time (PT) and activation partial thrombin time (APTT) ≤ 1.5×ULN; 10. Women of childbearing age must have a negative pregnancy test (βHCG) before starting treatment. Women of childbearing age and men (who have sex with women of childbearing age) must agree to use effective contraceptives continuously during treatment and 6 months after the last therapeutic dose; 11. Subjects signed the informed consent, and able to follow the planned visit, research treatment, laboratory examination and other experimental procedures.

Exclusion Criteria:

1. known as squamous carcinoma, undifferentiated cancer or other tissue types of gastric cancer, or adenocarcinoma mixed with other tissue types of gastric cancer;
2. HER2 positive stomach cancer patients: define IHC 3+, or IHC 2+ and FISH/ISH positive;
3. Previously received immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as antibodies to ICOS, CD40, CD137, GITR, OX40 targets, etc.) , immune cell therapy and other treatment of any immune mechanism for tumors;
4. In the first 14 days of randomization, there is still uncontrollable pleural hydration and ascites after puncture drainage and other treatments. Imaging shows that a small number of or medium chest and ascites patients can be selected for the study;
5. Subjects have not received prior systemic therapy for locally advanced or metastatic gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction. For subjects who have received prior neoadjuvant/adjuvant chemotherapy or chemoradiotherapy for curative intent, the time between disease progression and last treatment should be at least 6 months;
6. There are significant clinical bleeding symptoms or clear bleeding tendencies within 1 month before the first administration, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis;
7. There are clinically active hemoptysis, active diverticulitis, abdominal abscess, and gastrointestinal obstruction;
8. Any other malignant tumors have been diagnosed within 5 years before entering the study, except for skin basal or squamous cell carcinoma, superficial bladder cancer, cervical insitus, intraductal cancer and thyroid papilloma cancer that can be treated locally and have been cured with clear medical records;
9. Known active or untreated brain metastases, meningeal metastases, spinal cord compression, or leptomeningeal disease. However, subjects who meet the following requirements and have measurable lesions outside the central nervous system are allowed to enter the group: after treatment, the imaging is stable for at least 4 weeks before the start of the study treatment (if there is no new or expanded brain metastasis), and systemic glucocortic hormone and anticonvulsive drug treatment has been stopped at least 2 weeks;
10. Interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (such as diabetes, hypertension, pulmonary fibrosis and acute pneumonia, etc.) are known, and a history of active tuberculosis is known;
11. Subjects with active, known or suspected autoimmune disease. But Subjects who are in a stable state and do not require systematic immunosuppressive treatment are allowed, such as type 1 diabetes, hypothyroidism that only needs hormone replacement therapy, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or hair loss);
12. There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) NYHA level 2 and above cardiac insufficiency or cardiac ultrasound examination: LVEF (left ventricular ejection fraction) <50%; (2) severe/unstable angina pectoris; (3) randomized myocardial infarction within 6 months ; (4) Clinically significant supventricular or ventricular arrhythmia requires treatment or intervention; (5) Symptomatic congestive heart failure; (6) QTc>480 ms (QTc interval is calculated in the Fridericia formula; if QTc is abnormal, it can be separated by 2 minutes. The clock is detected 3 times in a row and takes its average value);
13. Received the following treatments or drugs before the first administration:

    1. Excessive surgery within the first 28 days (tissue biopsy required for diagnosis and peripheral vein puncture central venous catheterization [PICC] / infusion port implantation are allowed);
    2. Immunosuppressive drugs have been used within the first 14 days, excluding nasal spray and inhalation corticosteroids or systemic steroid hormones at physiological doses (i.e. no more than 10 mg/d prednisone or other corticosteroids of the same physiological dose of the drug);
    3. Inoculated with live attenuated vaccine within the first 28 days or within 60 days after the study period and the end of the research drug treatment;
    4. Receive local anti-tumor treatment within the first 28 days (such as radiotherapy or tumor embolization, etc.);
    5. Received Chinese herbal medicine or Chinese medicine with anti-tumor indications in the first 2 weeks;
14. Known allergies or intolerant to test drugs or their excipients; or a known history of severe hypersensitivity reactions to other monoclon antibodies;
15. Unable to swallow, malabsorption syndrome, or uncontrollable nausea, vomiting, diarrhea or other gastrointestinal diseases that seriously affect drug use and absorption;
16. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis (hepatitis B, defined as HBV-DNA≥500 IU/ml; hepatitis C, defined as anti-HCV positive and HCV RNA higher than analysis The lower limit of detection of the method) or combined with hepatitis B and hepatitis C;
17. Subjects who cannot comply with the test plan or cannot cooperate with the follow-up;
18. Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate,ORR | 6 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression free Survival | 1 year
  Defined as the time between signing the informed consent form to the disease progression (according to RECIST v1.1 criteria) or death due to any cause.
Overall survival | 2 years
  Defined as the time between signing the informed consent form to death due to various causes.
Disease Control Rate | 6 months
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1.
Duration of Response | 6 months
  Defined as the time from response(when CR or PR is first diagnosed) to disease progression or death due to any cause.
Incidence of adverse events | 6 months
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Overall Officials: yanqiao zhang, phD, Principal Investigator — Harbin Medical University Cancer Hosptital
Locations (1):
- Harbin Medical University Hospital, Harbin, China